CLINICAL TRIAL: NCT05443945
Title: Efficacy of ADW S-100 Ionized Water Nasal Spray in Decreasing Symptoms of Allergic Rhinitis: Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy of ADW S-100 Ionized Water Nasal Spray in Decreasing Symptoms of Allergic Rhinitis
Acronym: SPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P & B Group (Industry)
Collaborators: MediAxe CRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC2-2111.11NS
Record Dates: First submitted 2022-06-24; First posted 2022-07-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled study
  With a 4-7 days run-in period before a 14 days treatment/placebo period
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Water -100 ionized nasal spray (Experimental): 3 sprays in each nostril, 3 times a day during 14 days
  Interventions: Device: Nasal Spray
- Nasal spray with purified water (Placebo Comparator): 3 sprays in each nostril, 3 times a day during 14 days
  Interventions: Device: Nasal Spray

INTERVENTIONS:
Device: Nasal Spray — 3 sprays in each nostril 3 times per day

SUMMARY:
A nasal spray based on Advanced Water S-100 ionized water would clean the nasal cavities, reduce the viscosity of mucus and facilitate its elimination and decongestion of the nose and the prevention of the bridging of the allergen to the epithelial cells of the cavity nose at the origin of the onset of symptoms.

Indeed, a water-based nasal spray ionized Advanced Water S-100 would modify the electrostatic environment of all the interactions ensuring this bridging. Negative ions (OH-) contained in water ionized Advanced Water S-100 competes with negative ions from acids negatively charged amino acids and also neutralize basic amino acids positively charged. The destabilization of all the links governing the process of epitope/IgE association would prevent the bridging of the FcɛRI receptors of the mast cell and thus the cascade of cellular responses that cause symptoms.

The purpose of this study is to assess whether the use of ionized water nasal spray ADW S-100 allows to sufficiently reduce the intensity of the symptoms of allergic rhinitis and thus improve the quality of life of people with allergies.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years old
2. Inform consent
3. Beneficiaries of a social security scheme
4. Having documented persistent or intermittent allergic rhinitis for at least 2 years
5. In the respiratory environment allergen battery, at least one prick-test positive at selection (diameter >3mm compared to the negative control), or prick-test or specific IgE assay less than 6 months old demonstrating an allergic response appropriate
6. Agreeing not to take anti-allergic drug treatment during the duration of the study except in case of aggravation of the disease
7. Having a smartphone or a computer allowing access to the application of seizure

   To be eligible to be randomized, participants must have:
8. Used the nasal spray at least 2 times a day during the run-in, according to their answers on the application
9. A median VAS for the evaluation of the discomfort due to the symptoms of the selection at D-1 ≥ 50mm

Non-inclusion Criteria:

1. Existence of links with any member of the study staff or the sponsor, or conflicts interests with the promoter
2. Known hypersensitivity or allergy to one of the components of the product tested
3. Contraindication to the use of a nasal spray
4. Respiratory pathology other than allergic rhinitis/rhino-conjunctivitis and asthma mild or moderate. People with severe asthma may be included if their asthma is controlled
5. Current treatment with systemic corticosteroids
6. Known pregnancy or positive urine pregnancy test at screening and/or at D0, or breastfeeding in progress
7. Participation in a clinical trial or other clinical investigation using a device medicine for the treatment or prevention of rhinitis or conjunctivitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
percentage of patients with a change of at least 23 mm VAS (Visual Analogue Scale) at D4 | 14 days
  minimum 0 and maximum 100 (higher scores mean a worse outcome)

SECONDARY OUTCOMES:
percentage of change on D4 and D14 compared to D0 of symptoms (nasal obstruction, sneezing, rhinorrhea, sore throat) | 14 days
percentage of change on D4 and D14 compared to D0 of eye symptoms (itching, tearing, redness) | 14 days
VAS from D0 to D14 | 14 days
  minimum 0 and maximum 100 (higher scores mean a worse outcome)
Allergic rhinitis control test on D0 and D14 | 14 days
percentage of patients without symptoms at D4 and D14 | 14 days
percentage of patients who used antihistamines | 14 days
Proportion of premature discontinuations of the study or discontinuations of the product under study | 14 days
Proportion of attendees presenting events adverse events (AE), serious adverse events (SUE), AEs related to the product of the study, AEs of interest particular: respiratory infections | 14 days
Proportion of participants - satisfied or very satisfied - judging the use easy or very easy | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Lefevre, Dr, Principal Investigator — CHR Metz-Thionville
Locations (11):
- France (11):
  - GHEF, Jossigny, Seine Et Marne
  - CH Aix Maupertuis, Aix-en-Provence
  - CHR Metz-Thionville, Ars-Laquenexy
  - Cabinet Libéral, Lille
  - Hôpital Saint Vincent, Lille
  - Cabinet libéral, Manosque
  - Hôpital Nord - APHM, Marseille
  - CHU Montpellier, Montpellier
  - Centre d'allergologie de Gentilly, Nancy
  - Cabinet Libéral, Paris
  - Alyatec, Strasbourg